CLINICAL TRIAL: NCT00005788
Title: Phase II Trial of Subcutaneous Injections of Interleukin-2 for the Treatment of Mycosis Fungoides or the Sezary Syndrome
Brief Title: Interleukin-2 in Treating Patients With Mycosis Fungoides or Sezary Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low/inadequate rate of accrual.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 96H7; NU-96H7; NCI-G00-1735
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Lymphoma
Keywords: stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill lymphoma cells.

PURPOSE: Phase II trial to study the effectiveness of interleukin-2 in treating patients who have mycosis fungoides or Sezary syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with mycosis fungoides or Sezary syndrome treated with interleukin-2 (IL-2).
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive interleukin-2 subcutaneously for 4 consecutive days a week for 6 consecutive weeks. Treatment repeats every 8 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response or stable disease continue treatment for 2 courses past best response. Patients who demonstrate a persistent partial response continue treatment in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for survival.

PROJECTED ACCRUAL: A total of 15-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven mycosis fungoides or Sezary syndrome

  * Any stage
* Measurable disease with 1 or more indicator lesions

  * Evaluable disease for erythrodermic patients only
* At least 2 weeks since prior therapy, if documented progressive disease (PD)
* At least 4 weeks since prior therapy, if best response achieved without clear evidence of PD

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute granulocyte count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.2 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No cardiac pacemaker
* No clinically significant peripheral venous insufficiency

Other:

* No other malignancy within the past 5 years except:

  * Treated squamous cell or basal cell skin cancer
  * Treated carcinoma in situ of the cervix
  * Surgically treated other cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* HIV negative
* No poorly controlled diabetes mellitus

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* No concurrent steroids

Radiotherapy:

* See Disease Characteristics
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent proven or investigational antineoplastic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-04; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Kuzel, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (2):
- United States (2):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts